CLINICAL TRIAL: NCT03134365
Title: Factors to Determine the Responses to Meal Ingestion: Palatability
Brief Title: Palatability and Postprandial Sensations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PR(AG)338/2016C
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Healthy
Keywords: meal ingestion; palatability; postprandial responses; hedonic response

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mixed meal (Experimental)
  Interventions: Other: Mixed meal
- Combined meal (Active Comparator)
  Interventions: Other: Combined meal

INTERVENTIONS:
Other: Mixed meal — Mixed meal with identical composition and physical characteristics (colour, texture, consistency, temperature) but distinctively different palatability.
  Arms: Mixed meal
Other: Combined meal — Combined meal.
  Arms: Combined meal

SUMMARY:
Aim: to determine the effect of palatability on the cognitive (satiation/fullness) and emotive (digestive well-being/mood) responses to meal ingestion. The postprandial responses to conventional (potato and cheese cream followed by vanilla cream) versus unconventional test meals (mixture of both creams) with identical composition (350 Kcal) and physical characteristics (colour, texture, consistency, temperature) but distinctively different palatability will be studied on a cross over-design. The responses to the meals will be tested on 2 different days.

Participants (22 non-obese healthy men) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 5 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. Perception will be measured at 5 min intervals 10 min before and 20 min after ingestion and at 10 min intervals up to 60 min after the probe meal.

ELIGIBILITY:
Inclusion Criteria:

* non obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2016-11-23 (Actual); Study Completion 2016-12-02 (Actual)

PRIMARY OUTCOMES:
Meal palatability | 1 day
  Meal palatability measured by 10 score scales at the end of the test meal
Change in digestive well-being measured after the test meal | 1 day
  Change in average well-being measured by 10 score scales at the end of the test meal.

SECONDARY OUTCOMES:
Change in satiety measured after the test meal | 1 day
  Change in average satiety measured by 10 score scales at the end of the test meal
Change in fullness sensation measured after the test meal | 1 day
  Change in average fullness measured by 10 score scales at the end of the test meal
Change in abdominal discomfort/pain sensation measured after the test meal | 1 day
  Change in average abdominal discomfort/pain measured by 10 score scales at the end of the test meal
Change in mood measured after the test meal | 1 day
  Change in average mood measured by 10 score scales at the end of the test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain